CLINICAL TRIAL: NCT00824239
Title: Randomized Trial Comparing Intermittent Sedation and Daily Interruption of Sedation in Mechanically Ventilated Patients
Brief Title: Intermittent Sedation Versus Daily Interruption of Sedation in Mechanically Ventilated Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Antonio Paulo Nassar Junior, Antonio Paulo Nassar Junior, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0284/08
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Mechanical Ventilation
Keywords: critical care; sedation; Mechanically ventilated patients
MeSH Terms: interventions — Fentanyl; Midazolam; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Intermittent sedation (Active Comparator)
  Interventions: Procedure: Intermittent sedation
- 2. Daily interruption of sedation (Active Comparator)
  Interventions: Procedure: Daily interruption of sedation

INTERVENTIONS:
Procedure: Intermittent sedation — Patients under intermittent sedation stay without any continuous sedation since intubation and/or admission but receive analgesics as needed and sedatives only when agitated (SAS of 5 or more).
  Other Names: Fentanyl, midazolam, propofol
  Arms: 1. Intermittent sedation
Procedure: Daily interruption of sedation — Patients under daily interruption of sedation stay on continuous sedation with midazolam and fentanyl and are submitted to a daily interruption of sedation to a neurological evaluation until they reach a SAS of 4 or more, then continuous sedation is re-started in the half previous dosage.
  Other Names: Fentanyl, midazolam, propofol
  Arms: 2. Daily interruption of sedation

SUMMARY:
Sedation is very important in critical care. Critically ill patients are submitted to many stressor factors that have potential to affect longterm outcomes. However, oversedation is associated with increased morbidity, including increased time of mechanical ventilation and ICU stay and longterm psychological complications. Daily interruption of sedation is associated with less time under mechanical ventilation and less posttraumatic stress disorder. Intermittent sedation, when compared with continuous sedation, is also associated with decreased time of mechanical ventilation. The aim of this study is to compare intermittent sedation with daily interruption. Our primary endpoint is free-days of mechanical ventilation in 28 days.

DETAILED DESCRIPTION:
A comparison of intermittent sedation - keeping analgesia with fentanyl and midazolam or propofol as boluses if agitation (SAS 5 or more) after adequate analgesia - and daily interruption of sedation - analgesia with fentanyl and sedation wiht midazolam or propofol continuously with daily interruptions every morning until patients awake and can follow simple commands. Sedation is restarted in half previous dosage if agitation (SAS 5 or more) occur.

ELIGIBILITY:
Inclusion Criteria:

* Patients under mechanical ventilation with less of 24 hours and a expectative of stay intubated for more than 24 hours

Exclusion Criteria:

* Intubation secondary to a neurological cause
* Pregnant women
* Severe asthma or COPD decompensation
* Palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Ventilator free-days | 28 days

SECONDARY OUTCOMES:
Mortality | 28 days
Time of stay | ICU, hospitalar
Self-extubation | 28 days
Reintubation | 2 days after extubation
Incidence of posttraumatic stress disorder | 6 months
Unplanned withdrawal of catheters | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Paulo Nassar Junior, MD, Principal Investigator — University of Sao Paulo; Marcelo Park, PhD, Study Director — University of Sao Paulo
Locations (1):
- Hospital das Clinicas - University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Nassar Junior AP, Park M. Daily sedative interruption versus intermittent sedation in mechanically ventilated critically ill patients: a randomized trial. Ann Intensive Care. 2014 May 6;4:14. doi: 10.1186/2110-5820-4-14. eCollection 2014. PMID 24900938